CLINICAL TRIAL: NCT00023036
Title: Clinical and Molecular Analysis of Enlarged Vestibular Aqueducts
Brief Title: Clinical and Genetic Analysis of Enlarged Vestibular Aqueducts
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010228; 01-DC-0228
Record Dates: First submitted 2001-08-21; First posted 2001-08-22 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Sensorineural Hearing Loss; Cytomegalovirus Infection
Keywords: Genetics; Deafness; Genetic Markers; Genetic Analysis; GENETIC LINKAGE; Natural History; Hearing Impairment; Nonsyndromic Hereditary Hearing Impairment; SNHL; Inner Ear; Enlarged Vestibular Aqueducts; EVA
MeSH Terms: conditions — Hearing Loss, Sensorineural; Cytomegalovirus Infections; Deafness; Hearing Loss; Nonsyndromic sensorineural hearing loss

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Patients with known or suspected nonsyndromic SNHL associated with EVA
- 2: Patients with nonsyndromic EVA
- 3: unaffected siblings and parents of affected family members
- 4: Other unaffected relatives; included if there is more than one sibship with affected family

SUMMARY:
This study will try to identify and understand the genetic factors that lead to an inner ear malformation called "enlarged vestibular aqueducts", that can be associated with hearing loss.

Patients with sensorineural hearing loss with or without inner ear malformations and their parents and siblings may be eligible for this study. Participants and their immediate family members, may undergo some or all of the following tests and procedures:

* Medical and family history, including questions about hearing, balance and other ear-related issues, and review of medical records.
* Routine physical examination.
* Blood draw or buccal swab (brushing inside the cheek to collect cells) - Tissue is collected for DNA analysis to look for changes in genes that may be related to hearing loss.
* Hearing tests - The subject listens for tones emitted through a small earphone.
* Balance test (VEMP) to see if balance functions of the inner ear are associated with the hearing loss Electrodes will be placed behind your ear and at the base of your neck. From a reclining position, you will be asked to raise your head while clicking sounds are played into your ears. - Ultrasound tests - An inner ear malformation called EVA (enlargement of the vestibular aqueduct) indicates that a genetic disorder called Pendred syndrome may be the cause. Because thyroid abnormalities are also associated with Pendred syndrome, an ultrasound examination of the thyroid gland may be done.
* Computed tomography (CT) and magnetic resonance imaging (MRI) scans - These tests show the structure of the inner ear. For CT, the subject lies still for a short time while X-ray images are obtained. For MRI, the patient lies on a stretcher that is moved into a cylindrical machine with a strong magnetic field. The magnetic field and radio waves produce images of the inner ear. The radio waves cause loud thumping noises that can be muffled by the use of earplugs.

DETAILED DESCRIPTION:
Nonsyndromic hereditary hearing impairment is a genetically heterogeneous disorder that can be caused by mutations in any one of at least 60 different genes. Enlargement of the vestibular aqueduct (EVA) is a radiologic finding known to be associated with mutations in one of these genes, the Pendred syndrome gene (SLC26A4, formerly known as PDS). EVA may thus serve as a clinically useful marker to facilitate the diagnosis of hearing impairment. Recent data from our laboratory and others indicates that only a subset of individuals with EVA have SLC26A4 mutations, and therefore some EVA cases are likely to be caused by other genes, nongenetic factors, or a combination of these etiologies. Families with two or more individuals with hearing impairment and EVA will be enrolled in this study in order to identify other genetic factors that cause EVA. Siblings and parents may also be enrolled in order to define inheritance and to perform molecular genetic analyses.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must have or be a family member of a participant with known or non-syndromic SNHL associated with EVA or have evidence of other findings that suggest that EVA might be part of a novel phenotype

There must be at least two participating affected family members with one exception: if there is only one participating affected family member, there must be genetic test results identifying only one pathogenic mutant allele of SLC26A4

Adults must be able to provide informed consent

Minors must have a parent or guardian able to provide consent

Age between 0-99.

EXCLUSION CRITERIA:

Subjects with known exposure to physical or chemical teratogens in utero that could account for their inner ear malformations such as thalidomide or radiation

Any hearing loss that is associated with symptoms which meet the criteria of already known syndromes, such as, branchio-oto-renal (BOR) syndrome, which comprises system malformations and branchial cleft abnormalities and is caused by heterozygous mutations in the EYA1 gene.

Previous genetic testing identifying two pathogenic mutant alleles of SLC26A4.

Prospective study subjects who are cognitively impaired and lack consent capacity, will not be enrolled.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Affected and non-affected family members and affected single sporadic subjects with sensorineural hearing loss and enlarged vestibular aqueducts.
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2001-09-04 (Actual)

PRIMARY OUTCOMES:
By using genetic linkage, identify and map possible additional mutant alleles of SLC26A4 or other genes causing nonsyndromic EVA in patients with one or no detectable mutant allele of SLC26A4 | ongoing
  Identify genes other than SLC26A4 that cause EVA.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Friedman, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bauman NM, Kirby-Keyser LJ, Dolan KD, Wexler D, Gantz BJ, McCabe BF, Bale JF Jr. Mondini dysplasia and congenital cytomegalovirus infection. J Pediatr. 1994 Jan;124(1):71-8. doi: 10.1016/s0022-3476(94)70256-x. PMID 8283378
- [Background] Dahle AJ, Fowler KB, Wright JD, Boppana SB, Britt WJ, Pass RF. Longitudinal investigation of hearing disorders in children with congenital cytomegalovirus. J Am Acad Audiol. 2000 May;11(5):283-90. PMID 10821506
- [Background] Everett LA, Glaser B, Beck JC, Idol JR, Buchs A, Heyman M, Adawi F, Hazani E, Nassir E, Baxevanis AD, Sheffield VC, Green ED. Pendred syndrome is caused by mutations in a putative sulphate transporter gene (PDS). Nat Genet. 1997 Dec;17(4):411-22. doi: 10.1038/ng1297-411. PMID 9398842
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-DC-0228.html